CLINICAL TRIAL: NCT04384627
Title: Reducing Target Volumes in Patients With Locoregionally Advanced Nasopharyngeal Carcinoma Treated With Induction Chemotherapy Followed by Concurrent Chemoradiotherapy: A Phase 3, Multicentre, Non-inferiority, Randomised Controlled Trial
Brief Title: Reducing Target Volumes in NPC Treated With Induction Chemotherapy Followed by Concurrent Chemoradiotherapy
Acronym: NPC-GTV
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: First People's Hospital of Foshan (Other); Cancer Research Institute of Zhongshan City (Other Government)
Responsible Party: Principal Investigator, Ling-Long Tang, M.D., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5010-2019-09
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Nasopharyngeal Carcinoma; Induction Chemotherapy; Radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Intervention Model Description: Multicentre, Non-inferiority, Randomised controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pre-IC GTV (Active Comparator): The gross tumor volume (GTV) is delineated according to the pretreatment tumor extension
  Interventions: Radiation: Delineating the GTV according to the pretreatment or post-IC tumor extension
- Post-IC GTV (Experimental): The gross tumor volume (GTV) is delineated according to the post-IC tumor extension
  Interventions: Radiation: Delineating the GTV according to the pretreatment or post-IC tumor extension

INTERVENTIONS:
Radiation: Delineating the GTV according to the pretreatment or post-IC tumor extension — Delineating the GTV according to the pretreatment or post-IC tumor extension

SUMMARY:
To evaluate the long-term locoregional control, survival rate, late toxicity and quality of life after reducing the target volume in patients with locoregionally advanced nasopharyngeal carcinoma patients treated with induction chemotherapy plus concurrent chemoradiotherapy.

DETAILED DESCRIPTION:
This phase 3, multicenter, non-inferiority, randomized controlled clinical trial recruits patients with newly-diagnosed locoregionally advanced nasopharyngeal carcinoma patients treated with induction chemotherapy plus concurrent chemoradiotherapy. The intervention is delineating the gross tumor volume according to pretreatment tumor extension (the pre-IC GTV group) or post-induction chemotherapy tumor extension (the post-IC GTV group). The objective is to compare the long-term locoregional control, survival rate, late toxicity and quality of life between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* histologic confirmation of nonkeratinizing nasopharyngeal carcinoma; no previous treatment for cancer; nondistant metastatic, newly diagnosed stage III to IVa disease that was staged according to the American Joint Committee on Cancer-Union for International Cancer Control 8th edition stage-classification system; a Karnofsky performance-status score of at least 70 (on a scale from 0 to 100, with lower scores indicating greater disability); planned to receive 3 cycles of Induction Chemotherapy (regimens included docetaxel and cisplatin; docetaxel, cisplatin, and fluorouracil; and gemcitabine and cisplatin); and adequate hematologic, renal, and hepatic function.

Exclusion Criteria:

* younger than 18 years or elder than 70 years; receipt of treatment with palliative intent; a history of cancer; receipt of previous treatment (radiotherapy, chemotherapy, or surgery [except diagnostic procedures]) to the nasopharynx or neck; lactation or pregnancy; or severe coexisting illness; had disease progress after IC

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) | 3 year
  the time from randomization to documented locoregional recurrence or death from any cause

SECONDARY OUTCOMES:
Overall survival (OS) | 3 year
  the time from randomization to documented death from any cause
Late toxicities | 3 months
  Occur 3 months after IMRT, graded according to the Radiation Therapy Oncology Group radiation morbidity scoring criteria
Functional Assessment of Cancer Therapy-Head and Neck questionnaire (EORTC QLQ-H&N35) | 3 year
  Patient-reported QoL
Functional Assessment of Cancer Therapy-Head and Neck questionnaire (EORTC QLQ-C30) | 3 year
  Patient-reported QoL
Distant metastasis-free survival (DMFS) | 3 year
  DMFS was calculated from randomization to documented distant metastasis or death.
Acute toxicities | 3 months
  Occur within 3 months after IMRT

CONTACTS AND LOCATIONS:
Overall Officials: Ling-Long Tang, Principal Investigator — Sun Yat-sen University Cancer Centr
Locations (2):
- China (2):
  - First People's Hospital of Foshan, Foshan, Foshan
  - People's Hospital of Zhongshan City, Zhongshan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573
- [Background] Sun Y, Li WF, Chen NY, Zhang N, Hu GQ, Xie FY, Sun Y, Chen XZ, Li JG, Zhu XD, Hu CS, Xu XY, Chen YY, Hu WH, Guo L, Mo HY, Chen L, Mao YP, Sun R, Ai P, Liang SB, Long GX, Zheng BM, Feng XL, Gong XC, Li L, Shen CY, Xu JY, Guo Y, Chen YM, Zhang F, Lin L, Tang LL, Liu MZ, Ma J. Induction chemotherapy plus concurrent chemoradiotherapy versus concurrent chemoradiotherapy alone in locoregionally advanced nasopharyngeal carcinoma: a phase 3, multicentre, randomised controlled trial. Lancet Oncol. 2016 Nov;17(11):1509-1520. doi: 10.1016/S1470-2045(16)30410-7. Epub 2016 Sep 27. PMID 27686945
- [Background] Zhao C, Miao JJ, Hua YJ, Wang L, Han F, Lu LX, Xiao WW, Wu HJ, Zhu MY, Huang SM, Lin CG, Deng XW, Xie CH. Locoregional Control and Mild Late Toxicity After Reducing Target Volumes and Radiation Doses in Patients With Locoregionally Advanced Nasopharyngeal Carcinoma Treated With Induction Chemotherapy (IC) Followed by Concurrent Chemoradiotherapy: 10-Year Results of a Phase 2 Study. Int J Radiat Oncol Biol Phys. 2019 Jul 15;104(4):836-844. doi: 10.1016/j.ijrobp.2019.03.043. Epub 2019 Apr 5. PMID 30954521
- [Background] Yang H, Chen X, Lin S, Rong J, Yang M, Wen Q, Shang C, He L, Ren P, Xu S, Zhang J, Liu Q, Pang H, Shi X, Fan J, Sun X, Ma D, Tan B, Zhang T, Zhang L, Hu D, Du X, Zhang Y, Wen S, Zhang X, Wu J. Treatment outcomes after reduction of the target volume of intensity-modulated radiotherapy following induction chemotherapy in patients with locoregionally advanced nasopharyngeal carcinoma: A prospective, multi-center, randomized clinical trial. Radiother Oncol. 2018 Jan;126(1):37-42. doi: 10.1016/j.radonc.2017.07.020. Epub 2017 Aug 29. PMID 28864073
- [Background] McDowell LJ, Rock K, Xu W, Chan B, Waldron J, Lu L, Ezzat S, Pothier D, Bernstein LJ, So N, Huang SH, Giuliani M, Hope A, O'Sullivan B, Bratman SV, Cho J, Kim J, Jang R, Bayley A, Ringash J. Long-Term Late Toxicity, Quality of Life, and Emotional Distress in Patients With Nasopharyngeal Carcinoma Treated With Intensity Modulated Radiation Therapy. Int J Radiat Oncol Biol Phys. 2018 Oct 1;102(2):340-352. doi: 10.1016/j.ijrobp.2018.05.060. Epub 2018 Jun 4. PMID 30191868
- [Background] Sommat K, Ong WS, Hussain A, Soong YL, Tan T, Wee J, Fong KW. Thyroid V40 Predicts Primary Hypothyroidism After Intensity Modulated Radiation Therapy for Nasopharyngeal Carcinoma. Int J Radiat Oncol Biol Phys. 2017 Jul 1;98(3):574-580. doi: 10.1016/j.ijrobp.2017.03.007. Epub 2017 Mar 14. PMID 28581397
- [Derived] Tang LL, Chen L, Xu GQ, Zhang N, Huang CL, Li WF, Mao YP, Zhou GQ, Lei F, Chen LS, Huang SH, Chen L, Chen YP, Zhang Y, Liu X, Xu C, Zhao Y, Li JB, Liu N, Xie FY, Guo R, Sun Y, Ma J. Reduced-volume radiotherapy versus conventional-volume radiotherapy after induction chemotherapy in nasopharyngeal carcinoma: An open-label, noninferiority, multicenter, randomized phase 3 trial. CA Cancer J Clin. 2025 May-Jun;75(3):203-215. doi: 10.3322/caac.21881. Epub 2025 Feb 19. PMID 39970442